CLINICAL TRIAL: NCT01572285
Title: Transforaminal Epidural Steroid Injection to Treat Hemiplegic Shoulder Pain : A Randomized, Sham-Controlled, Proof of Principle Trial
Brief Title: Transforaminal Epidural Steroid Injection to Treat Hemiplegic Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0530/09
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-03

CONDITIONS: Hemiplegic Shoulder Pain
Keywords: Hemiplegic; Shoulder Pain; Transforaminal; Treatment; Interventional
MeSH Terms: conditions — Shoulder Pain | interventions — Dexamethasone; Steroids; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham (Sham Comparator): Sham arm received a simulation of transforaminal injection using a non-penetrating needle
  Interventions: Procedure: Sham
- Transforaminal (Experimental): Subjects received TF with infiltration of lidocaine 1% 0.5mL and 1.5mL of Dexamethasone 10mg/ml
  Interventions: Procedure: transforaminal dexamethasone injection

INTERVENTIONS:
Procedure: transforaminal dexamethasone injection — Subjects received transforaminal infiltration of lidocaine 1% 0.5mL and 1.5mL of Dexamethasone 10mg/ml
  Other Names: dexamethasone; steroid; transforaminal; TF; TFESI
  Arms: Transforaminal
Procedure: Sham — Sham procedure using a non-penetrating needle
  Arms: Sham

SUMMARY:
The purpose of this study is to determine whether transforaminal dexamethasone injections are effective in the treatment of chronic Hemiplegic Shoulder Pain.

DETAILED DESCRIPTION:
Shoulder pain is the most common complication in hemiplegia after Stroke (CVA). Almost three quarters of all patients with hemiplegia will suffer from shoulder pain in the first twelve months after stroke. Because of the lack of effective treatment today, the optimal management of hemiplegic shoulder pain is prevention. Although widely studied, all clinical trials for shoulder pain in stroke fail to show efficacy. TF was never investigated to treat Hemiplegic Shoulder Pain (HSP). The investigators hypothesize that injecting the epidural space at the C6 level via transforaminal would desensitize both central medullary components of pain as peripheral sensitized structures such as the suprascapular nerve of the affected shoulder.

To test this hypothesis, the investigators developed a treatment protocol consisting of two C6 transforaminal epidural steroid injection with dexamethasone (TF with 0.5mL of lidocaine 1% and 1.5mL of Dexamethasone 10mg/ml). This procedure was compared to a sham intervention.

ELIGIBILITY:
Inclusion Criteria:

* 3 months of shoulder pain following a stroke
* hemiplegia or paresis after a cerebral stroke for at least 6 months
* Shoulder pain greater than 4 in a visual analogue scale
* 50 to 65 years old

Exclusion Criteria:

* inability to understand or answer the tools in the study
* local inflammation or infection
* History of malignancy
* use of cardiac pacemaker
* allergy to lidocaine or dexamethasone
* disorders of coagulation

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-05 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Pain improvement after transforaminal injection using the Visual Analogue Scale (VAS) | 1 week and 3 months after treatment
  The primary outcome measures were pain measured using a visual analogue scale (VAS on a scale of 0≈10cm; where 0=no pain and 10=highest pain level during the last week).

SECONDARY OUTCOMES:
Algometry in shoulder muscles | 1 week and 3 months after treatment
  Algometry were measured in all shoulder muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Joao D Amadera, MD, Principal Investigator — University of São Paulo General Hospital
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil